CLINICAL TRIAL: NCT02780271
Title: Mi Vida Saludable: Maintaining Diet and Physical Activity Changes Among Latina Breast Cancer Survivors
Brief Title: Diet and Physical Activity Changes Among Latina Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dawn L. Hershman, Professor, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAP0461; R01CA186080 (NIH)
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cancer survivor; e-communication; diet and physical activity; fruits/vegetables daily servings; energy density
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Subjects will receive in-person education plus e-communication AND subjects will receive control intervention
  Interventions: Behavioral: In-person education; Behavioral: E-communication; Behavioral: Control
- Arm B (Experimental): Subjects will receive e-communication alone AND subjects will receive control intervention
  Interventions: Behavioral: E-communication; Behavioral: Control
- Arm C (Experimental): Subjects will receive in-person education alone AND subjects will receive control intervention
  Interventions: Behavioral: In-person education; Behavioral: Control
- Arm D (Active Comparator): Subjects will receive control intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: In-person education — Four in-person hands-on nutrition and physical activity education classes and cooking sessions.
  Arms: Arm A; Arm C
Behavioral: E-communication — 11 months of motivational text messages, emailed newsletters, and access to a website.
  Arms: Arm A; Arm B
Behavioral: Control — Written guidelines on diet and physical activity for breast cancer survivors, a pedometer to encourage physical activity, and a brief verbal overview of diet and physical activity guidelines for cancer survivors.

SUMMARY:
The investigators will conduct a 2x2 factorial randomized controlled trial to test the separate and synergistic effects of an in-person hands-on dietary and physical activity change curriculum (i.e., Mi Vida Saludable program) and e-communication strategies (text messaging, emailed newsletters and an interactive website) on changing dietary and physical activity behaviors among a diverse population of Latina breast cancer survivors who have completed breast cancer treatment. Participants will be evenly randomized to 4 arms: in-person education alone, e-communication alone, in-person education plus e-communication, or control.

DETAILED DESCRIPTION:
There are clear diet and physical activity guidelines for cancer survivors: eat a diet high in fruits/vegetables and low in energy-dense foods and engage in 150 minutes of moderate-to-vigorous physical activity each week. However, cancer survivors are provided with few, if any, resources to meet these guidelines and there are limited data supporting how cancer survivors can achieve sustained dietary change. There are even fewer behavioral change resources available to minority cancer survivors. Few studies have examined the separate and synergistic effects of in-person education and electronic or "e-"communication strategies in changing and maintaining health behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. 21 years of age or older.
3. Self-identify as Hispanic/Latina.
4. Speak Spanish or English.

   Disease Related Criteria
5. Medical history of histologically confirmed stage 0, I, II, III breast cancer, with no evidence of metastatic disease.

   Prior/ Current Therapy Criteria
6. At least 90 days post chemotherapy, biologic therapy, or radiation therapy treatment and/or breast surgery. Current use of hormonal therapy is permitted (e.g., tamoxifen and aromatase inhibitors).

   Accessibility Criteria
7. Have access to computer or smartphone.

   Clinical/ Laboratory Criteria
8. No history of smoking within the past 30 days.
9. No uncontrolled diabetes mellitus defined as Hgb A1C >7%
10. Consume <5 servings of fruits and vegetables per day and/or engages in <150 weekly minutes of moderate to vigorous physical activity.

Exclusion Criteria:

Any criterion not met under inclusion.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Change in daily servings of fruit/vegetables | Baseline, 6 months, 12 months
  Self-reported habitual fruit and vegetable intake will be assessed using the 10-item National Cancer Institute (NCI) All-Day Fruit and Vegetable screener.
Change in energy density | Baseline, 6 months, 12 months

SECONDARY OUTCOMES:
Change in Physical Activity | Baseline, 6 months, 12 months
  Physical activity will be measured using The International Physical Activity Questionnaire (IPAQ). The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marin-Chollom AM, Hale C, Koch P, Gaffney AO, Contento I, Shen H, Hershman DL, Brickman AM, Greenlee H. Cognitive Functioning and Health in Hispanic/Latina Breast Cancer Survivors. J Immigr Minor Health. 2022 Jun;24(3):597-604. doi: 10.1007/s10903-021-01300-w. Epub 2021 Oct 28. PMID 34709529
- [Derived] Santiago-Torres M, Contento I, Koch P, Tsai WY, Brickman AM, Gaffney AO, Thomson CA, Crane TE, Dominguez N, Sepulveda J, Marin-Chollom AM, Paul R, Shi Z, Ulanday KT, Hale C, Hershman D, Greenlee H. inverted exclamation markMi Vida Saludable! A randomized, controlled, 2 x 2 factorial trial of a diet and physical activity intervention among Latina breast cancer survivors: Study design and methods. Contemp Clin Trials. 2021 Nov;110:106524. doi: 10.1016/j.cct.2021.106524. Epub 2021 Aug 6. PMID 34365016